CLINICAL TRIAL: NCT02076581
Title: MyoSense- Automated Muscle Hypertonicity Classification System
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: The Cleveland Clinic (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: NS076052-1; 1R43NS076052-01A1 (NIH)
Record Dates: First submitted 2014-02-20; First posted 2014-03-03 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Stroke; Dystonia; Cerebral Palsy
MeSH Terms: conditions — Stroke; Dystonia; Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Stroke: Ten individuals with chronic stroke and limb spasticity will be recruited.
- Dystonia: Ten individuals with dystonic limbs and no spasticity will be recruited.
- Cerebral Palsy: Ten individuals with Cerebral palsy with the potential for a mix of dystonic and spastic abnormal tone in their affected limbs will be recruited.
- Neurologically normal: Thirty individuals without neurological injury that are age matched to the rest of the study population will be recruited.

SUMMARY:
It is often difficult to quantify and distinguish aspects of abnormal muscle tone due to neurological injury. This makes it difficult to evaluate therapies that aim to reduce the effects of abnormal muscle tone. This research study will evaluate the feasibility of a clinician worn device to capture and quantify features of spasticity and dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Presentation of dystonia and/or spasticity or, if in control group, no neurological injury nor abnormal muscle tone
* Over the age of five.

Exclusion Criteria:

* Intolerable pain with manipulation of the knee, ankle, wrist, or elbow
* Limited range of motion in the knee, ankle, wrist or elbow due to orthopedic injury or severe contraction.
* Cognitive impairment resulting in inability to provide informed consent or complete the protocol.
* Under the age of five.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sixty individuals, including individuals with and without abnormal muscle tone will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Correlation between clinician and device measured abnormal tone type. | For each subject clinician and device data will be collected within a single session. Each session will occur over a maximum of two hours. Analysis of all of the subject data will be completed within 30 days of study completion.
  Device measurements of clinician applied force relative to limb manipulation speed will be compared to conventional clinical outcome measures. For example, correlation between the slope of the force to speed profile and clinician evaluated spasticity, Ashworth score, will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Giuffrida, PhD, Principal Investigator — Great Lakes NeuroTechnologies Inc.
Locations (1):
- Great Lakes NeuroTechnologies, Valley View, Ohio, United States